CLINICAL TRIAL: NCT05996302
Title: Comparative Study of 6-minute Walk Distance (6MWD) in Patients With Pulmonary Vascular Diseases Permanently Residing Above 2500 Meters When Assessed Near Resident High Altitude (HA) at 2840m vs. at Low Altitude (LA) Sea Level.
Brief Title: HA Residents With PVD, 6MWD Assessed at HA (2840m) vs LA (Sea Level)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PVD_HAvsLA_6MWD
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Vascular Disease; Pulmonary Artery Hypertension; Chronic Thromboembolic Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Hypoxia; 6-minute walk test; High altitude; Pulmonary Artery Hypertension; Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Hypertension, Pulmonary; Hypoxia; Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Patients living permanently >2500m around Quito (Equador) will be assessed at 2850m and after relocation to sea level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-minute walk distance at 2840m (Active Comparator): Participants will have 6-minute walk distance (6MWD) assessment near their resident altitude at 2840m
  Interventions: Behavioral: Relocation to sea level
- 6-minute walk distance at sea level (Experimental): Participants will have 6-minute walk distance (6MWD) assessment at sea level (0-30m)
  Interventions: Behavioral: Relocation to sea level

INTERVENTIONS:
Behavioral: Relocation to sea level — Relocation to sea level by bus and stay for 2 days

SUMMARY:
To study the effect of relocation from 2840m (Quito) to sea level (Pedernales) in patients with pulmonary vascular diseases (PVD) defined as pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension (PH) who permanently live >2500m on 6-minute walk distance (6MWD)

DETAILED DESCRIPTION:
This research in patients with PVD diagnosed with precapillary PH with right heart catheterization and classified to groups 1 and 4 (PAH or CTEPH) who permanently live at HA >2500 (PVDHA) will have 6-minute walk distance near their living altitude in Quito at 2840m and at sea level in Pedernales the day after the first and the second night after relocation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-80 years old of both genders,
* Residence > 2500m of altitude
* diagnosed with precapillary PH (mean pulmonary artery pressure (mPAP) >20 mmHg, pulmonary artery wedge pressure (PAWP) ≤15 mmHg and pulmonary vascular resistance (PVR) ≥2 WU (wood units) by right heart catheterization) with PH being classified as PAH or CTEPH according to guidelines
* Patients stable on therapy
* NYHA (new york heart association) functional class I-III
* Provided written informed consent to participate in the study.

Exclusion Criteria:

* Age <18 years or >80 years
* unstable condition
* Patients who cannot follow the study investigations, patient permanently living < 2500m.
* Patients with moderate to severe concomitant lung disease (FEV1<70% or forced vital capacity <70%), severe parenchymal lung disease, severe smokers (>20 igarettes/day)
* Severely hypoxemic patients at Quito permanently have persistent SpO2 (oxygen saturation by pulseoximetry) <80% on ambient air.
* Patients with chronic mountain sickness (Hemoglobin > 19 g/dl in women, >21 g/dl in men)
* Patient with a non-corrected ventricular septum defect
* Relevant concomitant other disease of the heart, kidney, liver, blood (anemia hemoglobin<11 g/dl)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
6-minute walk distance (6MWD) after the first night at LA | after the first night at LA (sea level)
  Change in 6MWD in meter between LA (sea level) vs HA (2840 m)

SECONDARY OUTCOMES:
6-minute walk distance (6MWD) after the second night at LA | after the second night at LA (sea level)
  Change in 6MWD in meter between LA (sea level) vs HA (2840 m)
Arterial oxygen saturation by pulseoximetry (SpO2) at rest and at peak 6MWD after the first night at LA | after the first night at LA (sea level)
  Change in SpO2 in % between LA (sea level) vs HA (2840 m)
Arterial oxygen saturation by pulseoximetry (SpO2) at rest and at peak 6MWD after the second night at LA | after the second night at LA (sea level)
  Change in SpO2 in % between LA (sea level) vs HA (2840 m)
Heart rate at rest and at peak 6MWD after the first night at LA | after the first night at LA (sea level)
  Change in heart rate in bpm between LA (sea level) vs HA (2840 m)
Heart rate at rest and at peak 6MWD after the second night at LA | after the second night at LA (sea level)
  Change in heart rate in bpm between LA (sea level) vs HA (2840 m)
Blood pressure at rest and at peak 6MWD after the first night at LA | after the first night at LA (sea level)
  Change in blood pressure in mmHg between LA (sea level) vs HA (2840 m)
Blood pressure at rest and at peak 6MWD after the second night at LA | after the second night at LA (sea level)
  Change in blood pressure in mmHg between LA (sea level) vs HA (2840 m)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Departement of Pulmonology; Rodrigo Hoyos, Dr., Principal Investigator — Carlos Adrade Marin Hospital of Quito, Equador
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided upon request and based on a clear intention reviewed by an ethical review board.